CLINICAL TRIAL: NCT01312116
Title: Psychodynamic Versus Cognitive Behavioral Internet-Delivered Guided Self-help for Generalized Anxiety Disorder: A Randomized Controlled Trial
Brief Title: Psychodynamic Internet Treatment Versus Cognitive Behavioral Therapy (CBT) for Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Stockholm University (Other)
Responsible Party: Gerhard Andersson, Professor, Linköping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2007-0756
Record Dates: First submitted 2011-03-07; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: Internet treatment; GAD; guided self-help
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Internet-delivered CBT (Experimental): Active treatment: Internet-delivered Cognitive Behavior Therapy, 8 weeks treatment, guided self-help
  Interventions: Behavioral: iCBT
- Internet-delivered PDT (Experimental): Active treatment: Internet-delivered Psychodynamic Therapy Active treatment: Internet-delivered Psychodynamic Therapy, 8 weeks treatment, guided self-help
  Interventions: Behavioral: iPDT
- Control condition (No Intervention): Wait-list condition, received treatment 3 months after initial treatment period

INTERVENTIONS:
Behavioral: iCBT — Internet-delivered cognitive behavior therapy, 8 weeks
  Arms: Internet-delivered CBT
Behavioral: iPDT — Internet-delivered psychodynamic therapy, 8 weeks
  Arms: Internet-delivered PDT

SUMMARY:
The objective is to test if Internet-delivered cognitive behavior therapy (iCBT) or Internet-delivered psychodynamic therapy (iPDT) performs better for a population with generalized anxiety disorder (GAD), compared to a wait-list control condition.

DETAILED DESCRIPTION:
This was a non-inferiority trial within the context of a parallel group study with unrestricted randomisation in 1:1:1 ratio conducted in Sweden. Outcome assessors were blind to treatment status.

ELIGIBILITY:
Inclusion Criteria:

* fulfill the diagnostic criteria for GAD according to DSM-IV
* have access to the Internet
* have good knowledge of the Swedish language

Exclusion Criteria:

* recent (during last 6 weeks) change in psychiatric medication
* presently in any other psychological treatment
* severe depression
* suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | Two weeks pre treatment to two weeks post treatment.
  Change from baseline in anxiety symptoms to two weeks post treatment.

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale-Self Rated (MADRS-S) | Two weeks pre treatment to two weeks post treatment
  Change from baseline in depressive symptoms to two weeks post treatment.
Quality of Life Inventory (QOLI) | Two weeks pre treatment to two weeks post treatment
  Change from baseline in quality of life status to two weeks post treatment.
Beck Depression Inventory (BDI) | Two weeks pre treatment to two weeks post treatment
  Change from baseline in depressive symptoms to two weeks post treatment.
Beck Anxiety Inventory (BAI) | Two weeks pre treatment to two weeks post treatment
  Change from baseline in anxiety symptoms to two weeks post treatment.
Trimbos and iMTA questionnaire on Costs associated with Psychiatric illness (TIC-P) | Two weeks pre treatment to two weeks post treatment
  Change from baseline in societal cost of illness to two weeks post treatment.
State Trait Anxiety Inventory (STAI) | Two weeks pre treatment to two weeks post treatment
  Change from baseline in anxiety symptoms to two weeks post treatment.
Generalized Anxiety Disorder Questionnaire IV (GAD-Q IV) | Two weeks pre treatment to two weeks post treatment
  Change from baseline in anxiety symptoms to two weeks post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Professor, Study Director — Linkoeping University
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden

REFERENCES:
- See also: Project site — http://www.kbt.info/origo2/